CLINICAL TRIAL: NCT06904326
Title: Assessment of Spinal Stability by Dynamic Radiography After Unilateral Biportal Endoscopic Lumbar Decompression Surgery
Brief Title: CLUBE (UBE Stability / Dynamic Radio)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Principal Investigator, Guillaume LONJON, Principal Investigator, Clinique Saint Jean, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A00134-45
Record Dates: First submitted 2025-03-31; First posted 2025-04-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Spinal Instability
Keywords: biportal endoscopy; lumbar surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postoperative dynamic radiography (Experimental): all patients will perform a dynamic radiography 3 months after surgery
  Interventions: Other: Postoperative dynamic radiography

INTERVENTIONS:
Other: Postoperative dynamic radiography — Participants will perform a dynamic radiography 3 months after lumbar decompression surgery under UBE to study vertebral instability

SUMMARY:
Degenerative pathologies of the spine affect a large proportion of the increasingly ageing population, and are a major public health issue. When conservative treatments (physiotherapy, analgesics, infiltrations) fail, surgical treatment is preferred.

Traditionally, a simple lumbar recalibration operation is preferred (bilateral laminectomy decompression), but this may affect spinal stability. In cases of spondylolisthesis or preoperative instability, lumbar fusion (arthrodesis) is sometimes necessary to avoid the risk of major instability, but such an operation is not without risk and may require repeat surgery.

The development of new surgical techniques such as uni or bilateral laminotomies, which are less radical, has made it possible to avoid some arthrodeses. Nowadays, the emergence of new surgical techniques such as endoscopy has further reduced the risk of destabilization (shorter post-operative convalescence, less atrophy of the paraspinal muscles) and improved surgeon comfort (better vision and easier instrument handling).

Unilateral biportal endoscopy (UBE) is one of two endoscopic techniques and has proven its effectiveness for lumbar decompression in terms of clinical benefits. However, there is no scientific evidence on spinal stability after recalibration under UBE.

We believe that minimizing invasiveness with UBE during simple lumbar recalibration surgery can preserve spinal stability, thereby reducing the need for lumbar fixation and lowering the cost of care.

We therefore propose to study the maintenance of spinal stability using dynamic radiography at 3 months post-operatively in patients undergoing lumbar recalibration surgery with UBE.

DETAILED DESCRIPTION:
Spinal stability is defined by the absence of abnormal mobility (sagittal translation of at least 3 mm) between flexion and extension movements and will be assessed on the 3-months postoperative dynamic radiography.

Patients will undergone an additional dynamic radiography 3 months after surgery to assess their spinal stability.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 50 ans,
* Patient requiring single-level or 2-levels lumbar decompression surgery under UBE,
* Patients who underwent dynamic radiography within 3 months prior to surgery,
* Patient who received information on the study and who signed the consent form.

Exclusion Criteria:

* Presence of a mobile spondylolisthesis with a ≥ 3 mm difference between flexion and extension movements on preoperative dynamic radiography,
* Patient with history of lumbar arthrodesis,
* Patient not available for study follow-up.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Spinal stability rate | 3 months
  absence of abnormal vertebral mobility

SECONDARY OUTCOMES:
Spondylolisthesis rate | 3 months
Perioperative complications rate | 1 day
Oswestry Disability index evaluation | 3 months
  measure of patient incapacity improvement after surgery
Pain evaluation | 3 months
  measure of lumbar and radicular pain improvement after surgery with visual analog scale
Vertebral mobility evaluation | 3 months
  change in vertebral mobility between preoperative and postoperative dynamic radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique St Jean Sud de France, Montpellier, France

IPD SHARING:
Plan to Share IPD: No